CLINICAL TRIAL: NCT07384260
Title: The Effect of Probiotics on Gut Microbiota Changes in Healthy Chinese Adults During Short-Term European Travel: A Randomised, Double-Blind, Placebo-Controlled Clinical Trial
Acronym: The Effect of
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Min-Tze LIONG (Other)
Collaborators: Tsinghua University (Other)
Responsible Party: Sponsor-Investigator, Min-Tze LIONG, Prof., Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: THU-01-2025-1092
Record Dates: First submitted 2026-01-19; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Healthy Adult
Keywords: probiotic; international travel
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Daily 6-drops of non-GMO corn starch in medium-chain triglyceride oil
  Interventions: Other: Placebo
- Probiotic (Experimental): Daily 6-drops of Bifidobacterium animalis subsp. lactis B94, Lacticaseibacillus helveticus R0052 in non-GMO corn starch as excipient, in medium-chain triglyceride oil (1.5 × 109 CFU/day)
  Interventions: Other: Probiotic

INTERVENTIONS:
Other: Placebo — Daily 6-drops of non-GMO corn starch in medium-chain triglyceride oil
  Arms: Placebo
Other: Probiotic — Daily 6-drops of Bifidobacterium animalis subsp. lactis B94, Lacticaseibacillus helveticus R0052 in non-GMO corn starch as excipient, in medium-chain triglyceride oil (1.5 × 109 CFU/day)
  Arms: Probiotic

SUMMARY:
This study aims to evaluate the efficacy of a probiotic complex (containing Bifidobacterium animalis subsp. lactis B94 and Lacticaseibacillus helveticus R0052) in maintaining gut microbiota homeostasis and supporting physiological and psychological stability among healthy Chinese adults during short-term travel to Europe.

DETAILED DESCRIPTION:
With rising living standards, travel has become a common leisure activity. However, environmental changes, altered dietary habits, and disruptions to circadian rhythms during travel can significantly affect gut microbiota, potentially leading to various health issues. Dietary shifts are a primary driver of these alterations; the introduction of unfamiliar foods and beverages exposes the gut to foreign bacterial strains that compete with indigenous microbiota, increasing the risk of dysbiosis. This imbalance may manifest as gastrointestinal disturbances such as traveler's diarrhea or constipation, often associated with high-fat and low-fiber diets. In addition to dietary factors, travel-related stress, jet lag, and variations in hygiene conditions further influence microbial homeostasis. Growing evidence underscores a close relationship between gut microbiota and immune function, indicating that dysbiosis may compromise immune defenses and heighten susceptibility to respiratory infections and allergic responses triggered by novel environmental exposures.

Probiotics, defined as live microorganisms that confer health benefits when administered in adequate amounts, have gained considerable attention for their potential to promote human health. Predominantly derived from the *Lactobacillus* and *Bifidobacterium* genera, these beneficial microbes support gut health by modulating microbial composition, enhancing immune function, and improving digestive processes. Numerous studies have demonstrated their effectiveness in alleviating gastrointestinal disorders and reducing infection risk through immune system reinforcement. In addition, the capacity of probiotics to influence the gut-brain axis highlights their potential role in supporting mental health.

To ensure both safety and efficacy, this study employs *Bifidobacterium animalis* subsp. *lactis* B94 and *Lacticaseibacillus helveticus* R0052. Strain B94 has been clinically validated for improving bowel regularity and alleviating gastrointestinal discomfort through mechanisms such as short-chain fatty acid (SCFA) production, pathogen inhibition, and enhancement of intestinal barrier function. Strain R0052 is well recognized for its tolerability and its ability to shorten the duration of antibiotic-associated diarrhea while modulating immune responses. Moreover, R0052 has been shown to reduce psychological distress under stressful conditions, suggesting a regulatory role within the gut-brain axis. The combined use of these strains is therefore expected to promote microbiota stability and support overall health during the short-term physiological and psychological stress associated with travel.

The present study builds upon findings from a previous randomized controlled trial involving travelers to Japan. That trial demonstrated that short-term probiotic supplementation significantly enhanced gut microbiota resilience and improved both physiological and psychological homeostasis. Compared with the control group, participants receiving probiotics exhibited smaller fluctuations in microbial composition and achieved a more rapid return to baseline following travel. Lower incidences of gastrointestinal discomfort were reported, alongside improvements in anxiety, fatigue, and mood stability. Collectively, these results suggest that short-term probiotic intervention represents a practical and effective strategy for supporting health and well-being during periods of rapid environmental and lifestyle change.

ELIGIBILITY:
Inclusion criteria:

1. Aged 18-65 years, regardless of gender;
2. Planning to undertake a short-term round-trip journey to Europe (within 7 days);
3. Able to understand and willing to comply with the study protocol, and to cooperate with study procedures;
4. Voluntarily sign the informed consent form before any study-related procedures are initiated.

Exclusion criteria:

1. Diseases that may affect the evaluation of trial results, such as immune dysfunction, severe renal/hepatic dysfunction, severe cardiovascular disease, malignant tumors, acute or chronic infections, etc.;
2. Use of probiotic preparations, antibiotics, hormones, immunosuppressants, biological agents, or JAK inhibitors within 4 weeks;
3. Subjects with diagnosed or uncontrolled parasitic infections;
4. Patients receiving long-term medication for chronic diseases;
5. Patients with severe organic lesions in the thyroid, heart, brain, lungs, kidneys, or musculoskeletal system;
6. Patients with a history of or currently diagnosed mental illness;
7. Patients on long-term corticosteroid therapy;
8. Use of growth hormone, γ-aminobutyric acid (GABA), lysine, inositol, or vitamin B12;
9. Presence of uncontrolled, clinically significant laboratory abnormalities that may affect data interpretation or subject participation;
10. Participation in other clinical intervention studies involving drugs, dietary supplements, probiotics, or prebiotics within the past 4 weeks;
11. Presence of severe infections or major trauma deemed by the investigator to potentially affect outcomes, or having undergone moderate to major surgery within the past month;
12. Known allergy to any component of the probiotic product;
13. Subjects deemed unsuitable for participation by the investigator for any other reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Microbiota profiles of fecal samples in generally healthy adults upon administration of probiotic as assessed via metagenomics sequencing | 7 days
  Differences in microbiota abundance in fecal sample of generally healthy adults upon administration o probiotic compared to placebo

SECONDARY OUTCOMES:
Respiratory symptoms duration and frequency in generally healthy adults upon administration of probiotic as assessed using questionnaire | 7 days
  Changes in duration and frequency of respiratory illnesses symptoms from generally healthy adults on probiotic or placebo after 7-days, via the use of standard clinical assessment questionnaire, scale 0-3 where higher scores indicate more severe symptoms.
Gastrointestinal symptoms in generally healthy adults upon administration of probiotic as assessed using questionnaire | 7 days
  Differences in duration and frequency of gastrointestinal symptoms upon administration of probiotic compared to placebo via the use of standard clinical assessment questionnaire, scale 0-3 where higher scores indicate more severe symptoms.
Allergy symptoms in generally healthy adults upon administration of probiotic as assessed using questionnaire | 7 days
  Differences in duration and frequency of allergy symptoms upon administration of probiotic compared to placebo via the use of standard clinical assessment questionnaire, scale 0-3 where higher scores indicate more severe symptoms.
Anxiety in generally healthy adults upon administration of probiotic as assessed using questionnaire | 7 days
  Differences in anxiety using the Generalized Anxiety Disorder Scale (GAD-7), having a scale of 0-3 where higher scores indicate more severe outcomes, upon administration of probiotic compared to placebo.
Sleep quality in generally healthy adults upon administration of probiotic as assessed using questionnaire | 7 days
  Differences in sleep quality using the Pittsburgh Sleep Quality Index (PSQI), having a scale of 0-3 where higher scores indicate more severe outcomes, upon administration of probiotic compared to placebo.
General well being in generally healthy adults upon administration of probiotic as assessed using questionnaire | 7 days
  Differences in general well being using the World Health Organization Five Well-Being Index (WHO-5), having a scale of 0-5 where higher scores indicate better well being, upon administration of probiotic compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Ai Zhou, Ph.D., Principal Investigator — Tsinghua University Science and Technology
Locations (2):
- Tsinghua University Science and Technology, Haidian, Beijing Municipality, China
- Universiti Sains Malaysia, Pulau Pinang, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No